CLINICAL TRIAL: NCT04044833
Title: Evaluation of the Effects of Planned Trainings Given to Obese Adolescent Girls on Healthy Lifestyle Behaviors and Menstrual Symptoms:A Randomise Controlled Trial
Brief Title: Evaluation of the Effects of Planned Trainings Given to Obese Adolescent Girls on Healthy Lifestyle Behaviors and Menstrual Symptoms
Acronym: NuFaMeSTra
Status: Completed | Type: Observational
Sponsor: Hulya Erbaba (Other)
Responsible Party: Sponsor-Investigator, Hulya Erbaba, Ass. Prof. PhD., University of Beykent
Organization: University of Beykent (Other)
Other Study IDs: 521
Record Dates: First submitted 2019-07-29; First posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Obesity, Adolescent; Menstrual Problem; Health Behavior
MeSH Terms: conditions — Pediatric Obesity; Menstruation Disturbances; Health Behavior | interventions — Menstruation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- intervention: (n=63)
  Interventions: Behavioral: Health life style behaviour ,
- control: (n=65)
  Interventions: Behavioral: Health life style behaviour ,

INTERVENTIONS:
Behavioral: Health life style behaviour , — Training: applying Personal Information Form, HLBS-II, and MSQ to the intervention and control groups determined randomly and distributing the Student Follow-up Schedules; c) Providing trainings to the intervention group; d) Monitoring the weights, BMIs, and menstrual symptoms of intervention and control groups; and e) After the Training: Applying HLBS-II and MSQ scales to intervention and control groups, collecting the follow-up schedules, and providing training to the control group and all other students. Trainings: First stage: 120 minutes basic training per week for four weeks (40 minutes on diet, 40 minutes on physical activity, and 40 minutes on menstrual symptoms)
  Other Names: menstrual symptoms

SUMMARY:
The aim of this study is to evaluate the effects of training given to obese female students in mid-adolescence period for improving nutrition, physical activity, and menstrual symptoms on the improvement of their healthy lifestyle behaviors and menstrual symptoms. The research sample consisted of 128 obese female students divided into groups as intervention and control. In this randomized controlled trial, pretest-posttest control group and random process were used. In the first stage of the study, total of 12 hours of training, 120 minutes for each course per week, was provided. In the second stage, 120 minutes of reinforcement training were given every month for three months. The study lasted 16 weeks totally. Personal Information Form, Healthy Lifestyle Behavior Scale II (HLBS-II), Menstrual Symptom Questionnaire (MSQ) and Student Follow-up Schedule were used as data collection tools. Statistical analysis was performed using SPSS Statistics 23 Version. Hypotheses were (i) there was a difference between the total HLBS-II and MSQ scores of the students before and after the training and (ii) there was a correlation between the scales.

DETAILED DESCRIPTION:
Method The research was carried out as a randomized controlled trial to identify menstrual symptoms and healthy lifestyle behaviors of obese adolescent girls and to determine the effects of planned trainings given to them for improving nutrition, physical activity, and menstrual symptoms on the improvement of their healthy lifestyle behaviors and menstrual symptoms.

Research Hypotheses: H1: There is a difference between the mean scores of Healthy Lifestyle Behavior Scale II (HLBS-II) and H2: Menstrual Symptom Questionnaire (MSQ) before and after the trainings given to obese adolescent girls. H3: There is a correlation between the mean scores of HLBS-II and MSQ.

Study population and data collection tools: The study was carried out in three state high schools providing full-time education in a district of Ankara on September 1, 2017-January 21, 2018 and included 128 obese female students who accepted to participate voluntarily. These schools were chosen because the number of students was high and there were students from different socioeconomic levels. The study was approved by Yıldırım Beyazıt University Ethics Committee (decision numbered 12.04.2017/15 and coded 522). We obtained corporate permission from Ankara Provincial Directorate of National Education and informed consents of the students and their parents. Personal Information Form, HLBS-II, MSQ, and Student Follow-up Schedule, which were created by the researcher in accordance with the literature, were used as data collection tools.

Personal Information Form was prepared by examining the literature on the relevant age group to examine the demographic, nutritional, physical activity, and menstrual characteristics of the participants.10,11,14,16-19,22,23 Student Follow-up Schedule was developed for the students to record their menstrual pain and symptoms, weight and body mass index (BMI) measurements during the specified periods.

Menstrual Symptom Questionnaire was developed by Chesney and Tasto to assess menstrual pain and symptoms in 1975, and the usability of the questionnaire on adolescents was assessed by Negriff et al.24 and they updated the questionnaire in 2009. In 2013, Güvenç et al.24 conducted the reliability and validity study. Following the adaptation process, the questionnaire was prepared as 5-point Likert type and to involve 22 items. The MSQ score is calculated by taking the average of the total scores of the items in the scale. The increase in the mean score indicates that the severity of menstrual symptoms increases. The Cronbach's Alpha value of the scale is 0.86. In our study, it was found to be 0.91 and 0.92 before and after the trainings, respectively.

Healthy Lifestyle Behavior Scale II (HLSB-II): The scale was developed by Walker et al.25 in 1987 and updated in 1996 and named as Healthy Lifestyle Behavior Scale II. Bahar et al.26 studied the validity and reliability of its Turkish version in 2008. The 4-point Likert type scale consists of 52 items. Cronbach's Alpha value of the scale is 0.92. In our study, the Cronbach's Alpha value of the scale was found to be 0.91 and 0.92 before and after the trainings, respectively.

Treatment and control groups: The study population covers all female high school students. Study sample: In accordance with BMI-for-Age Percentile for Girls (kg/m2) determined by WHO,2 the study population was determined via two stages and consisted of volunteer female obese students aged 14 (BMI 26,7), 15 (BMI> 27,6) and 16 years (BMI> 28,2), who were currently at ninth, 10th and 11th grade in high school. In the first stage, BMIs, heights, and weights of 1300 female students who participated in the study voluntarily were measured and the students who met the criteria were included in the study. In the second stage, students, who agreed to participate in training and monitoring, were determined and they were, then, randomly divided into two groups, namely intervention (n=63) and control (n=65) groups.

The steps in the Implementation Phase are as follows: a) Sampling: measuring the BMIs, heights, and weights of 1300 female students, determining the sample group, and obtaining informed consent from them and their parents; b) Before the Training: applying Personal Information Form, HLBS-II, and MSQ to the intervention and control groups determined randomly and distributing the Student Follow-up Schedules; c) Providing trainings to the intervention group; d) Monitoring the weights, BMIs, and menstrual symptoms of intervention and control groups; and e) After the Training: Applying HLBS-II and MSQ scales to intervention and control groups, collecting the follow-up schedules, and providing training to the control group and all other students. Trainings: First stage: 120 minutes basic training per week for four weeks (40 minutes on diet, 40 minutes on physical activity, and 40 minutes on menstrual symptoms) . Second stage: Reinforcement trainings of 120 minutes were given once a month for three months. Periodic follow-up of intervention and control groups was carried out by recording their BMIs (Tanita BC 730 branded calibrated professional body analyzer was used to determine weight and BMI , which were measured three times in three periods) and menstrual symptoms ( participants were asked to mark Menstrual Pain and Symptoms in the first three days of menstruation in five periods) .

Statistical Analysis: Data was analyzed by using SPSS Statistics for Windows, Version 23.0 (IBM SPSS Statistics for Windows, Version 23.0. Armonk, NY: IBM Corp). Descriptive data was compared using Chi-Square and Mann-Whitney U tests, while Wilcoxon's and McNemar's tests were used to compare the menstruation findings of the students before and after the training. Dependent Samples t-Test was used in the intragroup comparison of total HLBS-II, MSQ, and sub-dimension scores. Comparison of differences between groups was performed by using the Independent Samples t-Test. Pearson's correlation analysis was used to determine the relationship between total HLBS-II and MSQ scores.

ELIGIBILITY:
Inclusion Criteria:

* Regular Menstruation
* Obese
* 9,10,11. class student

Exclusion Criteria:

Unregular menstruation non-attendance to training

Ages: 14 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — The research topic is menstrual symptoms and health life behaviours so we include girls as voluntary.
Study Population: : The study population covers all female high school students. Study sample: In accordance with BMI-for-Age Percentile for Girls (kg/m2) determined by WHO,2 the study population was determined via two stages and consisted of volunteer female obese students aged 14 (BMI 26,7), 15 (BMI> 27,6) and 16 years (BMI> 28,2), who were currently at ninth, 10th and 11th grade in high school. In the first stage, BMIs, heights, and weights of 1300 female students who participated in the study voluntarily were measured and the students who met the criteria were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-01-21 (Actual); Study Completion 2018-01-21 (Actual)

PRIMARY OUTCOMES:
Measurement of Health Life Style Behaviour Scale Points of Obese Adolescent Girls | 16 weeks
  Pretest intervention applied before to control and intervention groups. Nutrition, Physical Activity and Menstrual Symtoms Training given to intervention group (n=63) during the 16 weeks. After training posttest applied control and intervention groups. The health Life Style Behaviour Scale used for collect these data.
Measurement Menstruation Scale Points of Obese Adolescent Girls | 16 weeks
  Pretest intervention applied before to control and intervention groups. Nutrition, Physical Activity and Menstrual Symtoms Training given to intervention group (n=63) during the 16 weeks. After training posttest applied to control and intervention groups. The Menstruation Symptoms Scale used for collect these data.

SECONDARY OUTCOMES:
Measurements findings of menstruation pain according to the follow-up months of the students | 5 mounts
  The students menstruation pain followed up with a follow up form in control and intervention groups.

CONTACTS AND LOCATIONS:
Overall Officials: Hulya HE Erbaba, PhD, Principal Investigator — University of Beykent; sevil ss sahin, PhD, Study Director — UAnkara Yıldırım Beyazıt University
Locations (1):
- Kalaba Mesleki Teknik ve High School, Ankara, Kecıoren, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
I can send when they want
Supporting Information: Study Protocol
Time Frame: when they want I will send in a 30 day
Access Criteria: YÖKTEZ
URL: https://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp

DOCUMENTS (4):
  • Statistical Analysis Plan: Tables (2018-01-18): https://cdn.clinicaltrials.gov/large-docs/33/NCT04044833/SAP_000.pdf
  • Study Protocol: Consort Diagram and tables (2018-01-18): https://cdn.clinicaltrials.gov/large-docs/33/NCT04044833/Prot_001.pdf
  • Study Protocol: Consort (2018-01-18): https://cdn.clinicaltrials.gov/large-docs/33/NCT04044833/Prot_002.pdf
  • Statistical Analysis Plan: Tables (2018-01-18): https://cdn.clinicaltrials.gov/large-docs/33/NCT04044833/SAP_003.pdf